CLINICAL TRIAL: NCT03353961
Title: Internet Delivered Emotion Regulation Individual Therapy for Adolescents With Nonsuicidal Self-Injury: A Randomized Controlled Study
Brief Title: Internet Delivered ERITA for Nonsuicidal Self-Injury
Acronym: ERITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Clara Hellner Gumpert, PhD, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/10 BIP ERITA
Record Dates: First submitted 2017-11-02; First posted 2017-11-27 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Nonsuicidal Self-injury
Keywords: NSSI
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjunctive Internet-delivered ERITA (Experimental): Participants will receive 11 weeks of internet-delivered emotion regulation individual therapy with therapist support adjunctive to treatment as usual as provided in the community. The caregiver(s) will receive 6 modules of internet-delivered parent program with therapist support.
  Interventions: Behavioral: Emotion regulation individual therapy
- Treatment as usual (Active Comparator): Participants will receive treatment as usual for 11 weeks of treatment as usual as provided in the community.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Emotion regulation individual therapy — The emotion regulation individual therapy is delivered via an internet platform and includes therapist contact several times per week via the platform.
  Arms: Adjunctive Internet-delivered ERITA
Behavioral: Treatment as usual — Treatment as usual as provided in the community.
  Arms: Treatment as usual

SUMMARY:
To evaluate if Internet delivered emotion regulation individual therapy for adolescents is an efficacious treatment when delivered as adjunctive to treatment as usual compared to a control group consisting of treatment as usual.

DETAILED DESCRIPTION:
Statistical Analyses

Treatment effects will be evaluated according to the intention-to-treat principle. Primary end-point for all outcomes is post-treatment. Secondary end-point include a controlled 3 month follow-up.

Primary Analysis

The primary outcome analysis will include treatment group (ERITA , TAU) and weekly reports of NSSI frequency measured once every week 4 weeks prior to treatment start, once every week during treatment, and once every week four weeks after treatment termination. Regression analysis modelled for count data will be used to estimate trend over time. Four weeks after treatment termination will be considered primary endpoint. Pairwise contrasts (group x time interaction) from the regression model will be used to evaluate between-group differences at primary endpoint (4 weeks after treatment termination).

Secondary Analyses

Secondary outcomes measured once before, during, and after treatment will be analyzed in a similar fashion as for the primary outcome, modelled after data's distribution (count or continuous). Measures collected only once at baseline and post-treatment will be analyzed with regression analyses including treatment group (online ERITA , TAU) as the between-subjects factor, time (baseline to post) as the within-subjects factor, and group × time interactions, modelled after data's distribution (count or continuous).

Parallel process latent growth curve modeling will be used to determine whether change in week-to-week emotion dysregulation (DERS-16) during treatment mediate the overall effect of ERITA+ETAU on week-to-week change in the primary outcome self-rated NSSI frequency (DSHI-Y).

3 Month Follow-Up

Data collected at 3-month follow-up will be used to determine the extent to which potential treatment gains were maintained both within and between treatment conditions

Update 28 April 2022: As a secondary analyses, we also aim to investigate the effect of treatment moderators (primary aim) and predictors (secondary aim) on NSSI frequency one month after treatment termination. This update was submitted prior to conducting the analyses.

The selection of potential moderators was theoretically and empirically motivated. We will investigate the following variables (measured at baseline):

Age Difficulties in emotion regulation As measured with the Difficulties in Emotion Regulation Scale - 36 item version (DERS) Past month NSSI frequency As measured with the Deliberate Self-Harm Inventory Youth version (DSHI-Y) Global functioning As measured with the Childrens Global Assessment Scale Depressive symptoms As measured with the 21-item Depression Anxiety Stress Scales (DASS-21) Sleep difficulties As measured with the Insomnia Severity Index (ISI) Parental Minimization - discounting or devaluing the child's negative emotions/problems As measured with The Coping with Children's Negative Emotions Scale Adolescent Version (CCNES-A), subscale minimazation Level of suicidality As measured with the MINI-KID International Neuropsychiatric Interview, version 6

ELIGIBILITY:
Inclusion Criteria:

* ≥ 5 nonsuicidal self-injury episodes past year
* ≥ 1 nonsuicidal self-injury episodes past month
* having at least one parent who committed to participate in the parent program

Exclusion Criteria:

* Severe suicidal ideation
* a diagnosis of psychotic or bipolar I disorder or ongoing (past month) substance dependence
* the presence of co-occurring psychological disorders that required immediate treatment (i.e., severe anorexia nervosa)
* insufficient understanding of the Swedish language

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
Deliberate Self-Harm Inventory Youth version (DSHI-Y) | Change from baseline, once every week during treatment (0-12 weeks after baseline), 3 and 12 months after treatment has ended
  Frequency of nonsuicidal self-injury

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) | Change from baseline, once every week during treatment (0-12 weeks after baseline), 3 and 12 months after treatment has ended
  Difficulties in emotion regulation as primary potential mechanism of change. Ranges from 16-80, with higher scores indicating more difficulties.
Difficulties in Emotion Regulation Scale - 36 item version (DERS) | Change from baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
  Difficulties in emotion regulation. Ranges from 36-180, with higher scores indicating more difficulties.
the 21-item Depression Anxiety Stress Scales (DASS-21) | Change from baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
  Symptoms of depression, anxiety and stress. Each subscale (depression, anxiety and stress) ranges from 0-21, with higher scores indicating more symptoms.
Borderline Symptom List Supplement | Change from baseline, once every week during treatment (0-12 weeks after baseline), 3 and 12 months after treatment has ended
  Impulsive self-destructive behaviors
Acceptance and Action Questionnaire | Change from baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
  Acceptance and valued actions. Ranges from 7-49, with higher scores indicating less acceptance and valued actions.
Childrens Global Assessment Scale | Change from baseline, 16 weeks after treatment starts, 3 months after treatment has ended
  Global functioning. Ranges from 1-100, with higher scores indicating better functioning.
The Clinical Global Impressions -Severity and Improvement scales | Change from baseline, 16 weeks after treatment starts, 3 months after treatment has ended
  Global symptom severity and improvement. Severity of illness scale ranges from 1-7, with higher scores indicating higher severity of illness. Global improvement scale ranges from 1-7 with lower scores indicating more improvement.

OTHER OUTCOMES:
Short version of the Experiences in Close Relationships Scale - Revised Child version | Change from baseline, once every second week during treatment (0-12 weeks after baseline)
  Experiences in close relationships. Ranges from 12-84, with higher scores indicating greater problems.
Generalised Anxiety Disorder 7-item scale | Change from baseline, once every second week during treatment (0-12 weeks after baseline)
  Worry. Ranges 0-21, with higher scores indicating more worry.
Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness - Child version | Change from baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
  Costs associated with psychiatric illness
Kidscreen-10 | Change from baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
  Quality of life. Ranges 11-55, with higher scores indicating higher quality in life.
Patient Internet-delivered cognitive behavioral Adherence Scale | 6 and 12 weeks after baseline
  Patient adherence to treatment. Ranges from 0-20, with higher scores indicating higher adherence.
Working Alliance Inventory | 4 weeks after treatment starts
  Working alliance with online therapist
The Coping with Children's Negative Emotions Scale Adolescent Version | Change from baseline, 6 and 12 weeks after treatment starts, 3 and 12 months after treatment has ended
  Parents' perceived ability to cope with children's negative emotions. Three subscales will be used derived to reflect the specific types of coping response parents tend to use in these situations (punitive reactions, problem focused reactions, and minimization reactions). Each subscale ranges from 1-7.
The Client Satisfaction Questionnaire | 12 weeks after treatment starts
  Client satisfaction with treatment. Ranges from 8-32 with higher scores indicating greater treatment satisfaction.
Adverse Events | 12 weeks after treatment starts
  Self-rating scale that measures adverse events related to treatment
Credibility/Expectancy Questionnaire | 1 week after treatment starts
  Treatment credibility and expectancy. Ranges from 0-50 with higher scores indicating greater credibility/expectancy.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Hellner, PhD, MD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Centre for Psychiatry Research Karolinska Institutet and Stockholm County Council, Stockholm
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ojala O, Sjoblom K, Hesser H, Hedman-Lagerlof E, Hellner C, Bjureberg J. Parents' coping with their adolescent's negative emotions following internet-delivered emotion regulation therapy for adolescents with non-suicidal self-injury disorder: a secondary analysis of a randomised clinical trial. BMJ Ment Health. 2026 Jan 29;29(1):e302039. doi: 10.1136/bmjment-2025-302039. PMID 41611448
- [Derived] Ponten M, Flygare O, Bellander M, Karemyr M, Nilbrink J, Hellner C, Ojala O, Bjureberg J. Comparison between clinician and machine learning prediction in a randomized controlled trial for nonsuicidal self-injury. BMC Psychiatry. 2024 Dec 18;24(1):904. doi: 10.1186/s12888-024-06391-x. PMID 39695442
- [Derived] Bjureberg J, Ojala O, Hesser H, Habel H, Sahlin H, Gratz KL, Tull MT, Claesdotter Knutsson E, Hedman-Lagerlof E, Ljotsson B, Hellner C. Effect of Internet-Delivered Emotion Regulation Individual Therapy for Adolescents With Nonsuicidal Self-Injury Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2322069. doi: 10.1001/jamanetworkopen.2023.22069. PMID 37440232
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832